CLINICAL TRIAL: NCT05220137
Title: Using the Multiphase Optimization Strategy to Adapt Cognitive Processing Therapy
Acronym: CPT MOST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 21-088
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Stress Disorders, Post-Traumatic; Veterans; Psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Safety

STUDY DESIGN:
Intervention Model Description: Every condition in the experiment will begin with two initial core sessions (Rationale/Impact Statement and Working with Events, Thoughts, and Feelings) and end with a final core session. Each participant will then receive between one and five additional weekly sessions, as described below.
  The following CPT components will be empirically tested in the fractional factorial design: (1) Modified A-B-C, (2) Challenging Questions, (3) Patterns of Problematic Thinking, (4) Challenging Beliefs, and (5) Veteran's choice of Module (Safety/Trust/Power and Control/Esteem/Intimacy). Each component will be taught in a single session. As in standard CPT, each session will begin with a review of homework from the previous session, and then provide the listed component.
  All treatment sequences will end with a final session that consists of final homework review, review of treatment progress, and relapse prevention techniques. In total, participants will receive between 4 and 8 sessions.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (16):
- 1 (Active Comparator): Core Session 1, Core Session 2, Module Choice, Final Session
  Interventions: Behavioral: Veteran's choice of Module (Safety/Trust/Power and Control/Esteem/Intimacy)
- 2 (Active Comparator): Core Session 1, Core Session 2, Modified A-B-C, Final Session
  Interventions: Behavioral: Modified A-B-C: Working with Events, Thoughts, and Feelings
- 3 (Active Comparator): Core Session 1, Core Session 2, Challenging Questions, Final Session
  Interventions: Behavioral: Challenging Questions
- 4 (Active Comparator): Core Session 1, Core Session 2, Modified A-B-C, Challenging Questions, Module Choice, Final Session
  Interventions: Behavioral: Modified A-B-C: Working with Events, Thoughts, and Feelings; Behavioral: Challenging Questions; Behavioral: Veteran's choice of Module (Safety/Trust/Power and Control/Esteem/Intimacy)
- 5 (Active Comparator): Core Session 1, Core Session 2, Problematic Patterns, Final Session
  Interventions: Behavioral: Patterns of Problematic Thinking
- 6 (Active Comparator): Core Session 1, Core Session 2, Modified A-B-C, Problematic Patterns, Module Choice, Final Session
  Interventions: Behavioral: Modified A-B-C: Working with Events, Thoughts, and Feelings; Behavioral: Patterns of Problematic Thinking; Behavioral: Veteran's choice of Module (Safety/Trust/Power and Control/Esteem/Intimacy)
- 7 (Active Comparator): Core Session 1, Core Session 2, Challenging Questions, Problematic Patterns, Module Choice, Final Session
  Interventions: Behavioral: Challenging Questions; Behavioral: Patterns of Problematic Thinking; Behavioral: Veteran's choice of Module (Safety/Trust/Power and Control/Esteem/Intimacy)
- 8 (Active Comparator): Core Session 1, Core Session 2, Modified A-B-C, Challenging Questions, Problematic Patterns, Final Session
  Interventions: Behavioral: Modified A-B-C: Working with Events, Thoughts, and Feelings; Behavioral: Challenging Questions; Behavioral: Patterns of Problematic Thinking
- 9 (Active Comparator): Core Session 1, Core Session 2, Challenging Beliefs, Final Session
  Interventions: Behavioral: Challenging Beliefs
- 10 (Active Comparator): Core Session 1, Core Session 2, Modified A-B-C , Challenging Beliefs, Module Choice, Final Session
  Interventions: Behavioral: Modified A-B-C: Working with Events, Thoughts, and Feelings; Behavioral: Challenging Beliefs; Behavioral: Veteran's choice of Module (Safety/Trust/Power and Control/Esteem/Intimacy)
- 11 (Active Comparator): Core Session 1, Core Session 2, Challenging Questions, Challenging Beliefs, Module Choice, Final Session
  Interventions: Behavioral: Challenging Questions; Behavioral: Challenging Beliefs; Behavioral: Veteran's choice of Module (Safety/Trust/Power and Control/Esteem/Intimacy)
- 12 (Active Comparator): Core Session 1, Core Session 2, Modified A-B-C, Challenging Questions, Challenging Beliefs, Final Session
  Interventions: Behavioral: Modified A-B-C: Working with Events, Thoughts, and Feelings; Behavioral: Challenging Questions; Behavioral: Challenging Beliefs
- 13 (Active Comparator): Core Session 1, Core Session 2, Problematic Patterns, Challenging Beliefs, Module Choice, Final Session
  Interventions: Behavioral: Patterns of Problematic Thinking; Behavioral: Challenging Beliefs; Behavioral: Veteran's choice of Module (Safety/Trust/Power and Control/Esteem/Intimacy)
- 14 (Active Comparator): Core Session 1, Core Session 2, Modified A-B-C, Problematic Patterns, Challenging Beliefs, Final Session
  Interventions: Behavioral: Modified A-B-C: Working with Events, Thoughts, and Feelings; Behavioral: Patterns of Problematic Thinking; Behavioral: Challenging Beliefs
- 15 (Active Comparator): Core Session 1, Core Session 2, Challenging Questions, Problematic Patterns, Challenging Beliefs, Final Session
  Interventions: Behavioral: Challenging Questions; Behavioral: Patterns of Problematic Thinking; Behavioral: Challenging Beliefs
- 16 (Active Comparator): Core Session 1, Core Session 2, Modified A-B-C, Challenging Questions, Problematic Patterns, Challenging Beliefs, Module Choice, Final Session
  Interventions: Behavioral: Modified A-B-C: Working with Events, Thoughts, and Feelings; Behavioral: Challenging Questions; Behavioral: Patterns of Problematic Thinking; Behavioral: Challenging Beliefs; Behavioral: Veteran's choice of Module (Safety/Trust/Power and Control/Esteem/Intimacy)

INTERVENTIONS:
Behavioral: Modified A-B-C: Working with Events, Thoughts, and Feelings — The Modified A-B-C session teaches the Veteran how to draw connections between events, thoughts, and feelings and incorporates preliminary cognitive restructuring to help challenge stuck points. As in standard CPT, each session will begin with a review of homework from the previous session, and then provide the listed component.
  Arms: 10; 12; 14; 16; 2; 4; 6; 8
Behavioral: Challenging Questions — The Challenging Questions session teaches the Veteran to question and confront maladaptive self-statements and stuck points. As in standard CPT, each session will begin with a review of homework from the previous session, and then provide the listed component.
  Arms: 11; 12; 15; 16; 3; 4; 7; 8
Behavioral: Patterns of Problematic Thinking — The Patterns of Problematic Thinking session teaches the Veteran to identify counterproductive thinking patterns. As in standard CPT, each session will begin with a review of homework from the previous session, and then provide the listed component.
  Arms: 13; 14; 15; 16; 5; 6; 7; 8
Behavioral: Challenging Beliefs — The Challenging Beliefs session teaches the Veteran to generate alternative thoughts based on the outcome of cognitive restructuring. As in standard CPT, each session will begin with a review of homework from the previous session, and then provide the listed component.
  Arms: 10; 11; 12; 13; 14; 15; 16; 9
Behavioral: Veteran's choice of Module (Safety/Trust/Power and Control/Esteem/Intimacy) — The therapist will present the Module options to the Veteran and the Veteran will select one Module to work on. As in standard CPT, each session will begin with a review of homework from the previous session, and then provide the listed component.
  Arms: 1; 10; 11; 13; 16; 4; 6; 7

SUMMARY:
Cognitive Processing Therapy (CPT) consists of discrete therapeutic components that are delivered across 12 sessions, but most Veterans never reach session 12, and those who drop out receive only 4 sessions on average. Veterans drop out because of time constraints, logistics, and lack of perceived benefit. Unfortunately, Veterans who drop out prematurely may never receive the most effective components of CPT and continue to experience symptom-related distress and numerous other negative outcomes, including lost productivity, substance use, later-life physical disability, reduced quality of life, and increased risk of suicide.

The overall objective of this study is to adapt CPT into a brief, effective format. The rationale is that identifying the most effective intervention components and delivering only those components will make CPT deliverable in a shorter timeframe, thus improving efficiency, reducing drop-out related to poor treatment response, and ensuring that Veterans receive the most beneficial components of treatment, which will significantly improve their quality of life.

DETAILED DESCRIPTION:
Background: One third of post-9/11 Veterans in VHA suffer from posttraumatic stress disorder (PTSD), and among those who initiate Cognitive Processing Therapy (CPT), up to 70% drop out before receiving an adequate dose of treatment. Unfortunately, Veterans who drop out prematurely may never receive the most effective components of CPT. Thus, there is an urgent need to use empirical approaches to identify the most effective components of CPT, so that CPT can be adapted into a briefer format. The long-term goal of this line of research is to adapt, test, and implement brief, evidence-based treatment for Veterans with PTSD. The overall objective of the current application is to adapt CPT into a brief, effective format. The rationale is that identifying the most effective intervention components and delivering only those components will make CPT deliverable in a shorter timeframe, thus improving efficiency, reducing drop-out related to poor treatment response, and ensuring that Veterans receive the most beneficial components of treatment, which will significantly improve their quality of life.

Significance/Impact: Upon completion of this project, the investigators expect to have produced an empirically-based, brief version of CPT. This contribution is likely to improve clinical practice for Veterans with PTSD by providing the most effective components at an earlier session, thus increasing the overall effectiveness of treatment and mitigating the negative consequences of untreated PTSD, such as lost productivity, substance use, later-life physical disability, reduced quality of life, and increased risk of suicide. Using a highly efficient experimental design, we will identify which of five CPT components contribute meaningfully to reduction in PTSD symptoms. The investigators will test the effectiveness of each component and each two-way interaction between components.

Methodology: The MOST is an innovative engineering-inspired framework that uses an optimization trial to assess the performance of individual intervention components within a multicomponent intervention such as CPT. Guided by the MOST framework, the goal of the proposed project is to empirically inform an abbreviated version of CPT via a highly efficient fractional factorial design. Veterans (N = 270) at three VAMCs with clinically significant PTSD symptoms who meet minimal inclusion/exclusion criteria will be randomized to receive two or more CPT components. This design will test the effectiveness of each component and each two-way interaction between components, as measured by PTSD symptom reduction on the Clinician-administered PTSD scale for DSM-5 (CAPS-5) across six months of follow-up.

Implementation/Next Steps: Upon completion of these aims, the expected outcome is an adapted, abbreviated version of CPT that consists of the most effective elements of the intervention. The adapted intervention will be primed for a future large scale, fully powered effectiveness trial. The adapted intervention can be easily disseminated through the VA CPT training program and will have a positive impact on the health and wellbeing of Veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

The investigators designed the sample to be representative of Veterans with PTSD who are treated in PTSD Clinical Teams (PCTs), with minimal exclusion criteria. PCT clinicians will provide care for those with exclusionary comorbidities or preference for a medication-based approach, as per standard policies and procedures. Inclusion criteria are:

* score of 33 or above on the PCL-5
* at least 4 weeks on a stable dose for individuals who are taking psychotropic medication
* over the age of 18

Exclusion Criteria:

* active suicidality (assessed by the Columbia Suicide Severity Rating Scale with scores indicating elevated acute risk for suicide warranting hospitalization or intensive treatment)
* need for detoxification
* severe cognitive impairment that, in the judgment of the investigator, makes it unlikely that the patient can provide informed consent or adhere to the study regimen (as evidenced by confusion, inability to track discussion or answer questions, or other clear and significant indicators of cognitive impairment)
* psychosis or unmanaged bipolar disorder
* previous receipt of CPT in the past year
* current engagement in trauma-focused psychotherapy (Prolonged Exposure or Cognitive Processing Therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Change | Baseline, 6-week, 3-month, 6-month
  The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a 30-item structured interview used to measure of PTSD severity. In addition to assessing the 20 DSM-5 PTSD symptoms, questions target the onset and duration of symptoms, subjective distress, impact of symptoms on social and occupational functioning and improvement in symptoms since a previous CAPS administration.
  Scoring An index trauma/Criterion A event At least one Criterion B symptom (questions 1-5) At least one Criterion C symptom (questions 6-7) At least two Criterion D symptoms (questions 8-14) At least two Criterion E symptoms (questions 15-20) Both criterion F and G must be met as well for a PTSD diagnosis. To meet criteria for a symptom, a patient must meet criteria in both frequency and intensity score for each item. Frequency and intensity then combined to form a single severity score. Severity scores range from 0-4, with 0 being absent to 4 being extreme/incapacitating.

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) Change | Baseline, 6-week, 3-month, 6-month
  The PCL-5 is a 20-item self-report measure designed to assess PTSD symptoms as defined by the DSM-5. Each item of the PCL-5 is scored on a five point scale ranging from 0 ("not at all") to 4 ("extremely"). Items are summed to provide a total severity score (range = 0-80).The PCL-5 has strong internal consistency, test-retest reliability, and convergent and discriminant validity. Scores of 33 and above indicate a probable diagnosis of PTSD.
Patient Health Questionnaire (PHQ-9) Change | Baseline, 6-week, 3-month, 6-month
  The PHQ-9 is a 9-item self-report measure that assesses the presence and severity of depressive symptoms. Patients are asked to rate the presence of symptoms over the past 2 weeks on a 4-point likert scale ranging from 0-3 (not at all, several days, more than half the days, nearly every day) with a range of scores between 0-27. Total scores ranging from 5-9 indicate mild depression, 10-14 indicate moderate depression, 15-19 indicate moderately severe depression, and 20-27 indicate severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Kaufman Sripada, PhD MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (3):
- United States (3):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dodge J, Sullivan K, Grau PP, Chen C, Sripada R, Pfeiffer PN. Retention in Individual Trauma-Focused Treatment Following Family-Based Treatment Among US Veterans. JAMA Netw Open. 2023 Dec 1;6(12):e2349098. doi: 10.1001/jamanetworkopen.2023.49098. PMID 38127345
- [Result] Sripada RK, Peterson CL, Dziak JJ, Nahum-Shani I, Roberge EM, Martinson AA, Porter K, Grau P, Curtis D, McElroy S, Bryant S, Gracy I, Pryor C, Walters HM, Austin K, Ehlinger C, Sayer N, Wiltsey-Stirman S, Chard K. Using the multiphase optimization strategy to adapt cognitive processing therapy (CPT MOST): study protocol for a randomized controlled factorial experiment. Trials. 2023 Oct 19;24(1):676. doi: 10.1186/s13063-023-07669-3. PMID 37858262

DOCUMENTS (1):
  • Informed Consent Form (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT05220137/ICF_000.pdf